CLINICAL TRIAL: NCT07330141
Title: Optimizing Post-Chemotherapy Recovery: A Head-to-Head Trial of Graded vs. Constant-Load Aerobic Exercise in Pediatric ALL Survivors
Brief Title: Optimizing Recovery in Pediatric ALL Survivors: A Training Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT/0023/0029
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphobkastic Leukemia

STUDY DESIGN:
Intervention Model Description: A prospective, three-arm, randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: A single-blind protocol was adopted. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CL-AEx group (Experimental): The CL-AEx group received a 12-week constant-load aerobic training besides a structured exercise program.
  Interventions: Other: Constant-load Aerobic Exercise
- G-AEx group (Experimental): The G-AEx group received a 12-week intensity- and duration-graded aerobic training in addition to a structured exercise program.
  Interventions: Other: Graded Aerobic exercise
- Control group (Active Comparator): The control group received the structured exercise program only for 12 consecutive weeks.
  Interventions: Other: Structured Exercise regemin

INTERVENTIONS:
Other: Constant-load Aerobic Exercise — The CL-AEx group completed a 12-week, moderate-intensity aerobic training program in addition to the structured exercise regimen. The aerobic component was performed three times per week at a fixed intensity of 65% of the maximum age-predicted heart rate for 45 minutes per session. Each session included a 5-minute warm-up and a 5-minute cool-down. The intensity and duration remained constant throughout the intervention period.
  Arms: CL-AEx group
Other: Graded Aerobic exercise — The G-AEx group completed a 12-week aerobic training program that progressively increased in intensity and duration, in addition to the structured exercise regimen. Sessions were conducted three times per week. The program commenced at an intensity of 50% of the maximum age-predicted heart rate for 25 minutes. Parameters were increased every two weeks, culminating in an intensity of 75% for 50 minutes during the final two weeks. Each session included a standard 5-minute warm-up and 5-minute cool-down.
  Arms: G-AEx group
Other: Structured Exercise regemin — The structured exercise regimen was conducted three times per week for 45 minutes per session over 12 consecutive weeks. Each session consisted of flexibility exercises, progressive resistance training, balance training, and low-intensity conditioning activities.
  Arms: Control group

SUMMARY:
This study compared the effects of constant-load aerobic exercise (CL-AEx) and graded aerobic exercise (G-AEx) on cardiopulmonary fitness and functional capacity in pediatric survivors of acute lymphoblastic leukemia (ALL).

A cohort of 72 pediatric ALL survivors was randomly assigned to one of three groups: a CL-AEx group (n=24), a G-AEx group (n=24), or a control group (n=24). All groups participated in a structured exercise regimen. The CL-AEx group performed additional moderate-intensity aerobic training at a fixed load, while the G-AEx group performed additional aerobic training with progressive increases in intensity and duration. The control group performed the structured exercise regimen only. Interventions were administered three times per week for 12 consecutive weeks.

Cardiopulmonary fitness and functional capacity were assessed in all three groups at baseline and following the completion of the 12-week intervention.

DETAILED DESCRIPTION:
Seventy-two pediatric ALL survivors were recruited from the Pediatric Oncology and Hematology departments of three referral hospitals in the Riyadh region, Saudi Arabia. Inclusion criteria required participants to be aged 10-18 years, have completed chemotherapy, present with secondary sarcopenia, and possess normal cardiac structure and function without lower limb deformities. Participants were also required to be non-regular exercisers. Exclusion criteria included a history of secondary cancers, neurodegenerative impairments affecting memory, attention, or executive function, or any neuromusculoskeletal condition likely to impede training compliance (e.g., recurrent intensive cramps or impaired proprioceptive function).

Outcome Measures

Cardiopulmonary Fitness: Peak oxygen uptake (VO₂ peak) was assessed using the McMaster cycle ergometer protocol.

Functional Capacity: This was evaluated via three performance-based tests: the 6-Minute Walk Test (6MWT), the Timed Up and Down Stairs Test (TUDS), and the 4x10 Meter Shuttle Run Test.

Interventions

All interventions were delivered three times per week for 12 consecutive weeks under close supervision by an experienced pediatric physical therapist.

Constant-Load Aerobic Exercise (CL-AEx) Group: This group (n=24) performed a structured exercise regimen plus a moderate-intensity aerobic training program. The aerobic component was maintained at a constant intensity of 65% of the maximum age-predicted heart rate for 45 minutes per session, each preceded by a 5-minute warm-up and followed by a 5-minute cool-down.

Graded Aerobic Exercise (G-AEx) Group: This group (n=24) performed the same structured exercise regimen plus an aerobic program with progressive intensity and duration. Starting at 50% of maximum age-predicted heart rate for 25 minutes, the parameters were increased every two weeks, culminating at 75% for 50 minutes in the final two weeks. Each session also included a 5-minute warm-up and cool-down.

Control Group: This group (n=24) performed only the structured exercise regimen for 45 minutes per session. The regimen included flexibility exercises, progressive resistance training, balance training, and conditioning activities.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 and 18 years old
* Complete maintenance chemotherapy
* Normal cardiac structure and function
* Absence of lower limb deformities
* Not engaging in regular exercise regimens

Exclusion Criteria:

* Secondary cancers
* Neurodegenerative impairments affecting memory, attention, or executive functioning
* Neuro-musculoskeletal conditions are likely to impede the training.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2023-12-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | 2 months
  The peak oxygen uptake (mL/kg/min) was assessed through a symptom-free exercise tolerance test (i.e., the McMaster cycling protocol).

SECONDARY OUTCOMES:
Six-minute walk test | 2 months
  This test identified the maximum distance (m) that each patient was able to cover over six minutes on a straight flat 30-m walkway, without running or jogging. Walking is regarded as more efficient in line with a longer distance coverage.
4x10 meter Shuttle Run test | 2 months
  This test identified the maximum distance (m) that each patient was able to cover over six minutes on a straight flat 30-m walkway, without running or jogging. Walking is regarded as more efficient in line with a longer distance coverage.
Timed up and down stairs test | 2 months
  This test measured the time (seconds) that each patient took to climb up and down a 14-step stair flight (each 20 cm in height). Better performance is indicated by a shorter time.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No